CLINICAL TRIAL: NCT07296536
Title: Expert Consensus on the Use of Isotretinoin in Rejuvenation: A Delphi Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Venus Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: Isotretinoin-Rejuvenation
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Isotretinoin; Isotretinoin Adverse Reaction; Rejuvenation
Keywords: isotretinoin; rejuvenation; consensus; delphi method; Expert pannel

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Expert Panel: A cohort of dermatology and aesthetic medicine experts participating in a Modified Delphi process to develop consensus recommendations on Isotretinoin in Rejuvenation.

SUMMARY:
This expert consensus project explores the role of low-dose isotretinoin as a rejuvenative and preventive strategy for photoaging and sebaceous-driven skin changes. While isotretinoin is traditionally used for acne, increasing clinical experience suggests that carefully selected micro-dose and low-dose regimens may improve skin texture, pore size, sebaceous activity, and overall skin quality, with potential benefits in skin aging and maintenance rejuvenation programs.

DETAILED DESCRIPTION:
This study is a non-interventional, Delphi-based expert consensus project designed to establish recommendations for the use of isotretinoin in skin rejuvenation. While isotretinoin is primarily indicated for acne, accumulating clinical evidence and practitioner experience suggest that low-dose or micro-dose regimens may contribute to improvements in skin texture, fine lines, pore size, sebaceous activity, and overall skin quality. However, standardized guidance on indications, dosing, treatment duration, monitoring, and safety precautions is limited.

A panel of expert dermatologists with practical experience in isotretinoin therapy and skin rejuvenation will be invited to participate in multiple iterative Delphi rounds. Experts will rate agreement with proposed statements using a structured Likert scale. After each round, anonymized feedback will be provided, and statements not reaching consensus will be revised and re-evaluated until stable agreement is achieved.

The final output will consist of consensus-based recommendations reflecting practical, safe, and evidence-informed guidance for dermatologists considering isotretinoin for rejuvenation purposes. The study will also identify areas of uncertainty where further research is needed, supporting the safe expansion of isotretinoin applications beyond acne management.

ELIGIBILITY:
Inclusion Criteria:

* Board-certified dermatologists or equivalent.

  * 5 years clinical experience in dermatology.

Practical experience prescribing isotretinoin, including low- or micro-dose regimens for rejuvenation or acne.

Active engagement in clinical dermatology, teaching, research, or guideline development.

Willingness to participate in all Delphi rounds and provide informed consent.

Exclusion Criteria:

* Non-dermatology specialists.

Less than 5 years of clinical experience.

Lack of relevant isotretinoin experience.

Significant undisclosed conflict of interest with isotretinoin manufacturers.

Inability to participate in all Delphi rounds.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Target panel: 20-35 experienced dermatologists with practical knowledge of isotretinoin use for rejuvenation or acne.
  Recruitment: Purposive sampling, stratified to ensure diversity in:
  Practice setting (academic, private, public)
  Geographic location
  Years of experience
  Baseline data collected: Age, sex, region, practice setting, years of experience, isotretinoin prescribing frequency, research or guideline involvement, declared conflicts of interest.
  Panel retention strategy: Over-recruit by 10-20% to compensate for attrition; maintain anonymity of responses; clear instructions and timelines for participation.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 6-12 weeks
  Level of expert consensus on statements regarding the use of isotretinoin for skin rejuvenation, measured as the proportion of panelists reaching a predefined agreement threshold (e.g., ≥70-80%) per statement.

SECONDARY OUTCOMES:
Secondary Outcome | 6-12 weeks
  Consensus on patient selection criteria for rejuvenative isotretinoin.
  Consensus on dosing strategies (micro-dose, low-dose, cumulative dose, treatment duration).
  Consensus on monitoring protocols (clinical and laboratory).
  Consensus on safety measures, including pregnancy prevention and management of adverse effects.
  Consensus on integration with other rejuvenation therapies (topicals, procedures, photoprotection).
  Identification of areas without consensus, highlighting knowledge gaps and research priorities.

CONTACTS AND LOCATIONS:
Locations (1):
- Venus Research Center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Delphi studies do not collect patient data, medical records, biological samples, or identifiable clinical information. Experts only give opinions, not "IPD." Their responses are anonymized, and sharing identifiable expert-level responses is not required and often discouraged